CLINICAL TRIAL: NCT00188123
Title: Rapid Diagnosis of Myocardial Damage and Coronary Stenosis With MRI
Brief Title: Rapid Diagnosis of Myocardial Damage and Coronary Stenosis With Magnetic Resonance Imaging (MRI)
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Jonkoping County Hospital (Other); Medical Research Council of Southeast Sweden (Other Government)
Responsible Party: Linkoping universitet, Linkoping universitet
Other Study IDs: 151:2004/8333 MPA Sweden
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2005-09

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; MRI late enhancement; Atrial fibrillation
MeSH Terms: conditions — Myocardial Infarction; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis is that single-shot imaging of myocardial infarction is possible in atrial fibrillation using MRI late enhancement technique

DETAILED DESCRIPTION:
50 outpatients in Jonkoping County with a diagnosis of in-hospital myocardial infarction, are asked to participate in this study comparing segmented true FISP late enhancement with single-shot trueFISP late enhancement for the diagnosis of myocardial damage. The study does not intervene regarding treatment but is a comparison of the diagnostic power of the two MRI techniques.

ELIGIBILITY:
Inclusion Criteria:

in-hospital diagnosis of myocardial infarction

Exclusion Criteria:

pacemaker, not willing to participate, metallic objects in brain or eyes,

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an in-hospital diagnosis of myocardial infarction having permanent atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2005-09 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan E Engvall, MD, PhD, Principal Investigator — University Hospital, Linkoeping
Locations (1):
- Varnamo Hospital, Värnamo, Sweden